CLINICAL TRIAL: NCT06798909
Title: Kidney Transplant Preemptive Therapy or Prophylaxis (KPoP) for CMV Prevention in D+R- Recipients
Brief Title: Kidney Transplant Preemptive Therapy or Prophylaxis for CMV Prevention in D+R Recipients
Acronym: KPoP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00020695; 1R01AI184205-01 (NIH)
Record Dates: First submitted 2025-01-17; First posted 2025-01-29 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Cytomegalovirus (CMV); Kidney Transplant; Complications; Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-emptive Therapy (Experimental): 900 mg of Valganciclovir given orally twice daily to Preemptive Therapy subjects upon detection of CMV viremia until plasma PCR is negative on two consecutive weekly PCR test. All dosages adjusted for renal dysfunction.
  Interventions: Drug: Valganciclovir (Pre-emptive CMV Therapy)
- Prophylaxis (Active Comparator): 900 mg of Valganciclovir given orally once daily to subjects for 200 days post transplantation. All dosages adjusted for renal dysfunction.
  Interventions: Drug: Valganciclovir CMV Prophylaxis

INTERVENTIONS:
Drug: Valganciclovir (Pre-emptive CMV Therapy) — Valganciclovir, 900 mg given orally twice daily to Preemptive Therapy group subjects as a PET only after a positive CMV PCR test and stopped after PCR is negative for 2 consecutive weeks.
  Arms: Pre-emptive Therapy
Drug: Valganciclovir CMV Prophylaxis — Valganciclovir, 900 mg given orally once daily to all Prophylaxis group subjects for 200 days post transplantation as prophylaxis.
  Arms: Prophylaxis

SUMMARY:
This is a prospective, randomized multicenter trial of preemptive therapy (PET) vs. antiviral prophylaxis (AP) for prevention of cytomegalovirus (CMV) disease in adult D+R- kidney transplant recipients (KTR). Patients meeting study eligibility criteria and who have provided informed consent will be randomized (1:1) within 7 days of transplant to receive, in an open label design, either AP with valganciclovir 900 mg orally once daily or letermovir 480 mg orally once daily [both dose adjusted per Food and Drug Administration (FDA) label] for 200 days post-transplant), or PET (central lab weekly plasma polymerase chain reaction (PCR) monitoring for CMV deoxyribonucleic acidemia (DNAemia)) for 100 days post-transplant, with oral valganciclovir 900mg orally twice daily (or renally dosed per FDA label) at onset of CMV DNAemia at any level and continued until plasma CMV DNAemia is negative or below the level of quantitation in two consecutive weekly plasma samples. Study participants will be followed for pre-specified outcomes (clinical, laboratory, immunologic, safety) until withdrawal, death, or study closure, up to a maximum of 5.5 years post-transplant. Approximately 360 participants (180 participants in each group) will be randomized into the study.

Estimated Time to Complete Enrollment: 4 years

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legally authorized representative has provided written informed consent.
2. Age ≥ 18 years of age at the time of informed consent.
3. Negative for antibody to CMV as assessed in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory between 28 days prior to transplant and 7 days post-transplant, but prior to enrollment, and no history of positive CMV serology Immunoglobulin G (IgG) antibody
4. Received a first kidney transplant from a CMV seropositive donor in the past 7 days prior to enrollment
5. Individuals of reproductive (childbearing) potential must have a negative pregnancy test (serum or urine) collected prior to randomization (standard of care (SOC) results within 7 days prior to transplant may be used), and must also agree to use a medically approved method of contraception. Acceptable methods include: barrier method, intrauterine device (hormonal or non-hormonal), oral hormonal contraceptives, abstinence from the time of enrollment through 1 month after discontinuation of either PET or AP.

   NOTE: Individuals of reproductive potential are defined as individuals who have reached menarche and who have not been post-menopausal for at least 12 consecutive months with follicle stimulating hormone (FSH) ≥40 IU/mL or 24 consecutive months if an FSH is not available, i.e., who have had menses within the preceding 24 months, and have not undergone a sterilization procedure (e.g., hysterectomy, bilateral oophorectomy, or salpingectomy).
6. If male, and not surgically sterile, must agree to practice barrier method of contraception or abstinence from the time of enrollment through 1 month after discontinuation of either PET or AP.

Exclusion Criteria:

1. In the opinion of the investigator, participants who are unable or unwilling to undergo preemptive therapy protocol (weekly CMV PCR, etc.)
2. Patients who are breastfeeding or planning to breastfeed within 6 months post-transplant
3. Allergy to valganciclovir/ganciclovir or Letermovir
4. Receipt of immunoglobulin or CMV-specific immunoglobulin within the last 3 months (this includes COVID convalescent plasma)
5. Currently enrolled in another interventional study that, in the investigator's opinion, could affect evaluation of the safety and/or efficacy outcomes
6. Most recent platelet count post-transplant <25,000/uL
7. Most recent ANC performed post-transplant <1000/uL
8. Multi-organ transplant or have undergone prior organ transplant
9. Baseline immunodeficiency prior to transplant:

   1. Known or suspected human immunodeficiency virus (HIV) infection
   2. Congenital or acquired immunodeficiency
10. Unacceptable immunosuppression

    1. Receipt of desensitization therapy prior to kidney transplant, or
    2. Receipt of a blood type A, B, or O-incompatible kidney transplant, or
    3. Receipt or planned receipt of any of the following: belatacept, alemtuzumab, or rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of endpoint committee (EC)-confirmed CMV disease (either syndrome or end-organ) by 1-year post-transplant. | Within 1-year post-transplant

SECONDARY OUTCOMES:
Non-inferiority of PET (within a 10% margin) vs AP for EC-confirmed CMV disease by 1-year post-transplant, contingent on failure to meet the primary superiority endpoint. | by 1-year post-transplant
  Although the study sample size is powered to detect the superiority of one preventive strategy compared to the other, it is possible that the two approaches may have similar efficacy with respect to prevention of CMV disease. Therefore, should there be insufficient evidence to conclude superiority of one of the approaches, a key Secondary Outcome is a non-inferiority assessment of preemptive therapy to prophylaxis, assuming a non-inferiority margin of 10%. This margin is based on what is known about the effectiveness of the two approaches as published in literature and the potential that the two strategies could be similarly efficacious in preventing CMV disease. The success rate for the prophylaxis group is estimated to be ~80% based on a systematic review and meta-analysis with hypothesized success rates for the preemptive group expected to be higher.
Proportion of participants with investigator-determined CMV disease | by 1-year post transplant
Time in days to biopsy-proven acute rejection (BIPAR) | From date of randomization until the date of BIPAR from any cause, assessed up to 5.5 years
Time in days to graft loss | From date of randomization until the date of graft loss from any cause, assessed up to 5.5 years
Time in days to death | From date of randomization until the date of death from any cause, assessed up to 5.5 years
Mean estimated glomerular filtration rate (eGFR) in mL/min/1.73m2 at 1, 2, 3, and 4-years post-transplant | 1, 2, 3, and 4-years post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit P. Limaye, MD, Principal Investigator — University of California, San Francisco
Locations (5):
- United States (5):
  - University of California, San Francisco School of Medicine, San Francisco, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Robert Wood Johnson Health Network Barnabas Health, Livingston, New Jersey
  - Medical College of Virginia Commonwealth, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Limaye AP, Budde K, Humar A, Vincenti F, Kuypers DRJ, Carroll RP, Stauffer N, Murata Y, Strizki JM, Teal VL, Gilbert CL, Haber BA. Letermovir vs Valganciclovir for Prophylaxis of Cytomegalovirus in High-Risk Kidney Transplant Recipients: A Randomized Clinical Trial. JAMA. 2023 Jul 3;330(1):33-42. doi: 10.1001/jama.2023.9106. PMID 37279999
- [Background] Kotton CN, Kumar D, Caliendo AM, Huprikar S, Chou S, Danziger-Isakov L, Humar A; The Transplantation Society International CMV Consensus Group. The Third International Consensus Guidelines on the Management of Cytomegalovirus in Solid-organ Transplantation. Transplantation. 2018 Jun;102(6):900-931. doi: 10.1097/TP.0000000000002191. PMID 29596116